CLINICAL TRIAL: NCT04686929
Title: The Efficacy and Safety of Subcutaneous Abatacept in the Prevention of Acute Graft-versus-host Disease After Haplo-identical Donor Hematopoietic Cell Transplantation
Brief Title: Abatacept s.c. for aGVHD Prevention in Haplo-HCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, CHEN Jia, M.D., The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SZ9102
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Abatacept; Acute-graft-versus-host Disease; Haplo-identical HCT; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): The participants in Cohort 1 will receive abatacept s.c
  Interventions: Drug: Abatacept s.c.

INTERVENTIONS:
Drug: Abatacept s.c. — subcutaneous abatacept: 250mg (d-1) , 125mg (d+5, +14, +21, +28, +35, +42, +49, +56) combined with CsA, MTX, MMF.

SUMMARY:
Acute graft-versus-host disease (aGVHD) is a potentially fatal complication after allogeneic hematopoietic cell transplantation (HCT), particularly for that with a HLA-mismatched donor. Abatacept has been demonstrated as a potent drug to reduce the risk of aGVHD, but the efficacy of subcutaneous form has yet been investigated. This trial is designed to preliminarily determin the efficacy and saftey of subcutaneous abatacept in the prevention of aGVHD after haplo-identical HCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age≧18 years
2. ECOG score 0-2 / Karnofsky score≧80
3. haplo-HCT is proposed
4. Conditioning with motified Bu/Cy+ATG regimen
5. Having the following hematologic malignancies with transplant indications:

   1. Acute leukemia
   2. Myelodysplastic syndrome
   3. Aggressive lymphoma
6. Expected survival ≥ 3 months
7. Written informed Consent can be acquired
8. Agree to use effective contraception

Exclusion Criteria:

1. With a history of allo-HCT previously
2. Allergic/intolerant to Abatacept
3. Contraindications to the use of Abatacept
4. HIV infection, or active HBV infection or HCV infection
5. Uncontrolled active infection
6. Vital organ function intolerated to transplantation
7. Other malignancies except for the following diseases: malignant tumors that have been cured for at least 3 years without active lesions; adequete treated non-melanoma skin cancer, malignant amygdala, and carcinoma in situ without active lesions
8. Evidence of complications or medical conditions that may interfere with research or put the subjects at serious risk, including but not limited to severe cardiovascular disease (e.g. New York Heart Association grade III or IV heart disease, myocardial infarction in the past 6 months, unstable arrhythmia or unstable angina) and/or severe lung disease (e.g. history of severe obstructive lung disease and symptomatic bronchospasm)
9. Pregnant and lactational women
10. Any life-threatening disease, medical condition, or organ dysfunction unfit for participants, or may interfere with the absorption or metabolism of Abatacept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of overt aGVHD | 100 days post-HCT
  The incidence of grade II-IV aGVHD post-transplantation

SECONDARY OUTCOMES:
Incidence of aGVHD | 100 days post-HCT
  The incidence of grade I-IV aGVHD post-transplantation
Incidence of severe aGVHD | 100 days post-HCT
  The incidence of grade III-IV aGVHD post-transplantation
Early transplant-related mortality | 100 days post-HCT
  The incidence of early transplant-related mortality
Relapse | 100 days post-HCT
  The incidence of relapse/progression of underlying disease

OTHER OUTCOMES:
Engraft failure | 100 days post-HCT
  Failed to engraft with donor cells
Blood cell recovery | 100 days post-HCT
  Neutrophil count recover to 1000/ul and platelet count recover to 20000/ul

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided